CLINICAL TRIAL: NCT06920264
Title: Effect of Tranexamic Acid (TXA) Administered Prior to Shoulder Arthroscopy on Postoperative Pain Medication Usage: A Randomized Controlled Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Louis Joint Replacement Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-12-1991
Record Dates: First submitted 2021-10-06; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: This Study Will Evaluate Whether TXA Reduces Pain
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients who receive TXA will exhibit less pain (Active Comparator): as measured by opioid consumption and VAS for the first 72 hours after surgery
  Interventions: Drug: Tranexamic acid
- Patients who receive placebo will have higher pain (Placebo Comparator): placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Tranexamic acid — A total of 150 participants will be enrolled and randomized 1:1 to receive either a standard dose of TXA (1000 mg) or an equivalent volume of placebo (normal saline, NS) at the time of surgery. .
  Arms: Patients who receive TXA will exhibit less pain
Other: placebo — saline
  Arms: Patients who receive placebo will have higher pain

SUMMARY:
To our knowledge, no studies examining the use of TXA after shoulder arthroscopy in an outpatient setting have been published. This study will evaluate whether TXA reduces pain as measured by opioid consumption and a visual analog scale for pain (VAS) for the first 72 hours after surgery. Secondary outcomes will examine whether patients were satisfied overall with their postoperative pain control, whether the time to first opioid use is increased, and whether the surgeon perceives improved surgical visualization in patients who received TXA. We will also examine the number of times pump pressure was increased during the procedure to improve visualization.

DETAILED DESCRIPTION:
We will conduct a double-blind, placebo-controlled randomized clinical trial (RCT) to assess if there is benefit to use of TXA in shoulder arthroscopy. The study will include patients scheduled for rotator cuff repair with or without concomitant procedures. Patients undergoing shoulder arthroscopy for any other reason will be excluded, including isolated labral repair, isolated distal clavicle excision, frozen shoulder, isolated decompression or debridement. Medical exclusion criteria will include allergy or known sensitivity to TXA, known renal disease with previously documented creatinine >1.5, history of coagulopathy, DVT or PE requiring ongoing anticoagulation, baseline long-acting opioid use, a documented history of COVID-19 infection within 90 days of surgery.

A total of 150 participants will be enrolled and randomized 1:1 to receive either a standard dose of TXA (1000 mg) or an equivalent volume of placebo (normal saline, NS) at the time of surgery. The primary outcome measure will be postoperative opioid consumption as measured by pill count for 72 hours, calculated as morphine equivalent dose (MED). Secondary outcome measures will include subjective measurement of pain as rated on the VAS, time to first opioid use, and patient satisfaction with postoperative pain management at 72 hours. Operative time, surgeon rating of overall visibility during the procedure, and number of times pump pressure was increased during the procedure will also be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to have shoulder arthroscopy with the PI (KAB)
* shoulder arthroscopy for partial or full thickness rotator cuff tear confirmed on MRI or CT arthrogram preoperatively.
* willing to sign consent to participation and randomization.

Exclusion Criteria:

* Surgical exclusion criteria:

  1. Revision procedures
  2. Irreparable tears including planned allograft augmentation and superior capsular reconstruction (SCR) procedures
  3. Goutallier staging for fatty infiltration of 3 or higher
  4. Substantial underlying arthritis (Samuelson and Prieto grade 2 or higher).

Medical exclusion criteria:

1. Allergy, known sensitivity to TXA.
2. Renal insufficiency as defined by serum creatinine >1.5 prior to surgery.
3. History of coagulopathy, DVT or PE requiring ongoing anticoagulation.
4. Baseline opioid use of long-acting medications including Fentanyl patches, Oxycontin CR, or MS Contin.
5. Documented history of COVID-19 infection within 90 days of surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-09-08 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
primary outcome measure will be postoperative opioid consumption as measured by pill count for 72 hours, calculated as morphine equivalent dose (MED). | 72 hours

SECONDARY OUTCOMES:
Secondary outcome measures will be postoperative pain management satisfaction at 72 hours. | 72 hours
  include VAS, time to first opioid use, and patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Burns, MD, Principal Investigator — SSM Health Orthopedics
Locations (1):
- SSM Health- DePaul, Bridgeton, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin ZX, Woolf SK. Safety, Efficacy, and Cost-effectiveness of Tranexamic Acid in Orthopedic Surgery. Orthopedics. 2016 Mar-Apr;39(2):119-30. doi: 10.3928/01477447-20160301-05. Epub 2016 Mar 4. PMID 26942474
- [Background] Pauzenberger L, Domej MA, Heuberer PR, Hexel M, Grieb A, Laky B, Blasl J, Anderl W. The effect of intravenous tranexamic acid on blood loss and early post-operative pain in total shoulder arthroplasty. Bone Joint J. 2017 Aug;99-B(8):1073-1079. doi: 10.1302/0301-620X.99B8.BJJ-2016-1205.R1. PMID 28768785
- [Background] Kirsch JM, Bedi A, Horner N, Wiater JM, Pauzenberger L, Koueiter DM, Miller BS, Bhandari M, Khan M. Tranexamic Acid in Shoulder Arthroplasty: A Systematic Review and Meta-Analysis. JBJS Rev. 2017 Sep;5(9):e3. doi: 10.2106/JBJS.RVW.17.00021. PMID 28902659
- [Background] Hurley ET, Lim Fat D, Pauzenberger L, Mullett H. Tranexamic acid for the Latarjet procedure: a randomized controlled trial. J Shoulder Elbow Surg. 2020 May;29(5):882-885. doi: 10.1016/j.jse.2020.01.066. PMID 32305106
- [Background] Liu YF, Hong CK, Hsu KL, Kuan FC, Chen Y, Yeh ML, Su WR. Intravenous Administration of Tranexamic Acid Significantly Improved Clarity of the Visual Field in Arthroscopic Shoulder Surgery. A Prospective, Double-Blind, and Randomized Controlled Trial. Arthroscopy. 2020 Mar;36(3):640-647. doi: 10.1016/j.arthro.2019.10.020. Epub 2019 Dec 20. PMID 31870749
- [Background] Karaaslan F, Karaoglu S, Yurdakul E. Reducing Intra-articular Hemarthrosis After Arthroscopic Anterior Cruciate Ligament Reconstruction by the Administration of Intravenous Tranexamic Acid: A Prospective, Randomized Controlled Trial. Am J Sports Med. 2015 Nov;43(11):2720-6. doi: 10.1177/0363546515599629. Epub 2015 Sep 2. PMID 26337246